CLINICAL TRIAL: NCT00033722
Title: A Phase II Multicenter Study Of Lometrexol Sodium And Folic Acid In Subjects With Previously Treated Stage IIIB or IV Non-Small Cell Lung Cancer
Brief Title: Lometrexol Plus Folic Acid in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tularik (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069316; TULA-T064031; USO-01103
Record Dates: First submitted 2002-04-09; First posted 2003-08-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2002-11

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Folic Acid; lometrexol

INTERVENTIONS:
Dietary Supplement: folic acid
Drug: lometrexol

SUMMARY:
RATIONALE: Lometrexol may stop or slow the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Folic acid may be effective in preventing or lessening the side effects of lometrexol. Combining lometrexol with folic acid may be an effective treatment for non-small cell lung cancer.

PURPOSE: Phase II trial to study the effectiveness of combining lometrexol with folic acid in treating patients who have stage IIIB or stage IV non-small cell lung cancer that has been previously treated.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall response rate in patients with previously treated stage IIIB or IV non-small cell lung cancer when treated with lometrexol and folic acid.
* Determine the complete response rate, duration of response, and time to progression in patients treated with this regimen.
* Determine the 1-year survival rate and overall survival in patients treated with this regimen.
* Determine the safety profile of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral folic acid once daily on days -7 to 6. Patients also receive lometrexol IV over 30-60 seconds on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed up to 2 months after removal from study and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 50-100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer (NSCLC)

  * Stage IIIB or IV

    * Squamous cell carcinoma
    * Adenocarcinoma
    * Large cell carcinoma
    * Adenosquamous carcinoma
* Progressive disease after receiving 1 cisplatin- or carboplatin-containing regimen for stage IIIB or IV disease
* Measurable disease

  * At least 1 lesion at least 1 cm x 1 cm by CT scan either not in a previously irradiated field or showing clear evidence of disease progression after radiation
* No symptomatic or rapidly increasing, moderate or large amounts of pleural effusion or ascites
* No prior or concurrent CNS metastases (brain or meningeal)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3*
* Platelet count at least 100,000/mm^3*
* Hemoglobin at least 9.0 g/dL*
* *Without transfusions or growth factors in the previous 7 days

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN) (regardless of liver involvement secondary to tumor)
* AST and ALT no greater than 2.5 times ULN (5 times ULN if liver has tumor involvement)

Renal:

* Calculated creatinine clearance at least 60 mL/min using Cockroft and Gault formula

Gastrointestinal:

* No inflammatory bowel disease
* No radiation enteritis
* No malabsorption syndrome
* No inability to absorb folic acid

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during study
* No known untreated vitamin B12 deficiency
* HIV negative
* No drug abusers
* No prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No severe concurrent disease or major comorbidity that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior biologic therapy for NSCLC and recovered from acute side effects
* Prior treatment with an experimental vaccine allowed
* No concurrent routine or prophylactic filgrastim (G-CSF), sargramostim (GM- CSF), or epoetin alfa

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy for NSCLC (6 weeks for mitomycin or nitrosourea) and recovered from acute side effects
* Prior adjuvant or neoadjuvant chemotherapy allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* Recovered from acute side effects of prior radiotherapy
* No prior radiotherapy to 25% or more of bone marrow
* No prior whole pelvic irradiation

Surgery:

* At least 3 weeks since prior major surgery and recovered

Other:

* At least 3 weeks since prior investigational agent
* No concurrent proguanil, trimethoprim, co-trimoxazole, or pyrimethamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-02

CONTACTS AND LOCATIONS:
Overall Officials: David Tesarowski, Study Chair — Tularik
Locations (7):
- United States (7):
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Cancer Centers of Florida (U.S. Oncology), Orlando, Florida
  - Louisiana State University School of Medicine, New Orleans, Louisiana
  - US Oncology - Albany Regional Cancer Center, Albany, New York
  - U.S. Oncology Research Inc., Houston, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Cancer Care Northwest, Spokane, Washington